CLINICAL TRIAL: NCT06763055
Title: The Fifth INTEnsive pReventing Secondary Injury in Acute Cerebral Haemorrhage Trial Within ACT-GLOBAL
Acronym: INTERACT5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ACT-GLOBAL_ICH_01
Record Dates: First submitted 2024-12-17; First posted 2025-01-08 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Intracerebral Hemorrhage; Spontaneous Intracerebral Hemorrhage; Supratentorial Intracerebral Haemorrhage; Acute Intracerebral Haemorrhage; Acute Stroke
Keywords: Stroke; Acute Stroke; ICH; Intracerebral Hemorrhage; Platform Trial; Adaptive Platform Trial; Supratentorial ICH; secondary brain injury; deferoxamine mesylate; colchicine
MeSH Terms: conditions — Cerebral Hemorrhage; Stroke | interventions — Colchicine; Deferoxamine

STUDY DESIGN:
Intervention Model Description: The INTERACT5 Domain includes two treatments provided in a factorial manner, creating four different treatment arms. The two treatments are: A. Intravenous deferoxamine mesylate (abbreviated as DX) B. Low-dose oral colchicine (abbreviated as OC)
  The four arms including three interventions and one control in the domain are the 2x2 factorial of each treatment/no treatment. The one control arm and three intervention arms in the domain are:
  1. No DX and No OC (labeled as Control)
  2. Yes DX and No OC
  3. No DX and Yes OC
  4. Yes DX and Yes OC
Who Masked: Outcomes Assessor
Masking Description: The trial will have allocation concealment and blinded endpoint assessment, but open-label treatment. Given the time sensitive nature of acute stroke treatment, blinding the enrolling personnel to treatment assignment is not practical. Clinical site staff, including the Principal Investigator (PI), sub-investigators, clinic site staff, and the Sponsor will not be blinded to treatment allocated or received. In the event of an emergency the PI will be already unblinded.
  The trial will have blinded endpoint assessment on Day 90, with central blinded assessors contacting the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No deferoxamine mesylate, No colchicine (control) (Placebo Comparator): The group will not receive deferoxamine mesylate or colchicine
  Interventions: Other: Control (Standard treatment)
- Deferoxamine mesylate only (Active Comparator): The intervention group will receive deferoxamine mesylate at a dose of 32mg/kg/day via intravenous infusion immediately (within 1 hour) of randomization and continued for 2 consecutive days.
  Interventions: Drug: Deferoxamine Mesylate
- Colchicine only (Active Comparator): The intervention group will receive 0.5mg of oral colchicine daily as soon as possible after randomization, to continue for 30 days.
  Interventions: Drug: Colchicine 0.5 mg
- Both deferoxamine mesylate and colchicine (Active Comparator): The intervention group will receive deferoxamine mesylate at a dose of 32mg/kg/day via intravenous infusion immediately (within 1 hour) and continued for 2 consecutive days; plus 0.5mg of oral colchicine daily as soon as possible after randomization, to continue for 30 days.
  Interventions: Drug: Colchicine 0.5 mg; Drug: Deferoxamine Mesylate

INTERVENTIONS:
Drug: Colchicine 0.5 mg — The intervention group will receive 0.5mg of oral colchicine daily as soon as possible after randomization, to continue for 30 days.
  Arms: Both deferoxamine mesylate and colchicine; Colchicine only
Drug: Deferoxamine Mesylate — The intervention group will receive deferoxamine mesylate at a dose of 32mg/kg/day via intravenous infusion immediately (within 1 hour) and continued for 2 consecutive days
  Other Names: Yes DX
  Arms: Both deferoxamine mesylate and colchicine; Deferoxamine mesylate only
Other: Control (Standard treatment) — The group will not receive deferoxamine mesylate or colchicine
  Arms: No deferoxamine mesylate, No colchicine (control)

SUMMARY:
This is a domain within the ACT-GLOBAL platform trial to compare the effectiveness of early and appropriate pharmacological interventions in acute intracerebral hemorrhage (ICH) to control secondary brain injury. Up to 2000 patients with presumed spontaneous supratentorial intracerebral hemorrhage (ICH) will be followed for 6 months (or death, if prior to 6 months).

Adaptive interim analyses will be used, with statistical triggers to determine if any of the interventions are superior to control. The end of the trial is defined as the date that all participants have completed their 6-month assessment.

A large amount of preclinical data indicates that the outcome from ICH is linked to the detrimental effects of breakdown substances from brain bleeds. However, there remains a lack of compelling evidence supporting the effectiveness of any pharmacological intervention that can mitigate the secondary cerebral injury. The INTERACT domain aims to assess the effectiveness of intravenous deferoxamine and low-dose oral colchicine, both individually and in combination, to standard of care alone, on improving functional outcome in patients with spontaneous supratentorial ICH.

Those patients who meet eligibility criteria will be randomized to receive one of four interventions:

1. No deferoxamine mesylate and no colchicine (labeled as control)
2. Deferoxamine mesylate only: deferoxamine mesylate at a dose of 32mg/kg/day via intravenous infusion immediately (within 1 hour) post-randomization and continue for the following 2 consecutive days.
3. Colchicine only: 0.5mg of oral colchicine daily for 30 consecutive days.
4. Both deferoxamine mesylate and colchicine: deferoxamine mesylate at a dose of 32mg/kg/day via intravenous infusion immediately (within 1 hour) post-randomization and continue for the following 2 consecutive days; plus 0.5mg of oral colchicine daily for 30 consecutive days.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) is a severe type of stroke, responsible for substantial disability and death worldwide. It accounts for 6.5% to 19.6% of all strokes, with incidence rates increasing, especially in low- and middle-income countries. Survivors often face significant consequences, including functional impairments, recurrent strokes, cognitive decline, and depression.

Despite advancements in acute stroke care, there are few effective treatments specifically targeting the brain damage caused by ICH. Previous research has identified that the formation of perihaematomal oedema (PHE) is a critical factor in poor recovery, making it a key focus for therapeutic development.

INTERACT5 domain will focus on two promising medications. Deferoxamine, an iron-chelating agent, targets oxidative stress caused by iron released from damaged brain tissue. Studies suggest it may reduce brain swelling and secondary injury after ICH. Colchicine, an anti-inflammatory medication, inhibits pathways involved in inflammation, which may help minimize brain damage. INTERACT5 will enroll patients aged 18-80 with acute spontaneous supratentorial ICH, confirmed through imaging, who present to the hospital within 24 hours of symptom onset. Other domain-specific inclusion criteria:

* Hematoma volume ≥≥10 mL or any volume post-surgery
* NIHSS score >8
* GCS ≥8>7

Participants will be randomized to one of four groups: standard care, deferoxamine alone, colchicine alone, or both treatments combined. Deferoxamine will be administered intravenously (32 mg/kg/day within 1 hour and continued for 2 consecutive days), and colchicine will be given orally (0.5 mg daily for 30 days).

The study's primary outcome is the improvements in functional outcomes at 6 months, measured by the modified Rankin Scale (mRS). Secondary outcomes include EQ-5D-5L at 6 months, changes in PHE size, NIHSS scores, length of hospital stay, ambulatory status at discharge and safety indicators such as mortality at 6 months/SAEs to 6 month, kidney and liver function.

Response Adaptive Randomization (RAR) will be used in this domain to allow readjustment of recruitment towards treatment arms with more favorable emerging effects. Randomization will use minimization method to minimize the imbalance between the number of patients in each treatment group over a number of factors including region, location (deep vs cortical)age (>65 vs ≤65 years old), sex (male vs female), time from onset (>6 vs ≤6 hours), haematoma volume (10-29 vs ≥30 mL), receipt of any decompressive surgery (yes vs no), and intraventricular extension of ICH, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years old
2. Diagnosis of presumed spontaneous supratentorial intracerebral haemorrhage, confirmed by brain imaging
3. Presentation to hospital within 24 hours of symptom onset (or last seen well)
4. Hematoma volume ≥10 mL or any volume post-surgery
5. NIHSS score >8
6. GCS ≥8
7. Provide written informed consent by patient (or approved surrogate)

Exclusion Criteria:

1. Secondary cause of haemorrhage (e.g., structural abnormality such as arteriovenous malformation, cerebral aneurysm, tumour, trauma), or haemorrhagic transformation of acute ischaemic stroke
2. Isolate intraventricular haemorrhage
3. Chronic Kidney Disease
4. Very high likelihood of death within 7 days or poor adherence to study treatment or follow-up
5. Severe comorbid disease that will interfere with outcome assessments (e.g., cancer, chronic airflow disease, heart failure, significant disability)
6. Women who are pregnant or lactating

   Exclusion Criteria related to use of deferoxamine:
7. Previous chelation therapy or known hypersensitivity to deferoxamine products;
8. Severe iron deficiency anaemia (haemoglobin <7 g/dL or requiring regular blood transfusions);
9. Taking iron supplements containing >325 mg of ferrous iron;
10. Serum creatinine >2 mg/dL;
11. Patients with known heart failure taking >500 mg of vitamin C

    Exclusion criteria related to the use of colchicine:
12. Allergic to colchicine
13. Myelodysplastic hypoplasia, or liver or severe renal failure
14. Use of medication which may interact with colchicine (e.g., strong CYPsA4 inhibitors such as ketoconazole, strong P-glycoprotein inhibitors such as fluconazole)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
mRS scores at 6 months analysed with utility-weights | From enrollment to the 6 month assessment
  Modified Rankin Scale (mRS) -which scores of 0 to 1 indicate a favorable outcome without or with symptoms but no disability, scores of 2 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.

SECONDARY OUTCOMES:
Excellent functional neurological outcome (mRS 0-1) at 6 months | From enrollment to the 6 month assessment
  Modified Rankin Scale (mRS) with scores of 0 to 1 indicating a favorable outcome without or with symptoms but no disability.
Independent functional neurological outcome (mRS 0-2) at 6 months | From enrollment to the 6 month assessment
  Modified Rankin Scale (mRS) with scores of 2 to 5 indicating increasing levels of disability (and dependency).
Health-related quality of life, as measured by the EQ-5D-5L at month 6 | Completed by telephone at the Day 90 assessment (Day 90 outcomes are assessed in a blinded manner)
  The EQ-5D-5L is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five response categories corresponding to: no problems, slight, moderate, severe and extreme problems. The version of the instrument selected for the trial is interviewer administered either in-person, or by telemedicine or by telephone. The respondents will also rate their overall health on the day of the interview on a 0-100 visual analogue scale (EQ-VAS).
Ordinal shift in the 7 levels of mRS at 6 months | Done at the 6-month assessment (assessed in a blinded manner)
  Modified Rankin Scale (mRS) in which scores of 0 to 1 indicate a favorable outcome without or with symptoms but no disability, scores of 2 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
Disability (mRS 3-5) at 6 months | Done at the 6-month assessment (assessed in a blinded manner)
  Modified Rankin Scale (mRS) in which scores of 0 to 1 indicate a favorable outcome without or with symptoms but no disability, scores of 2 to 5 indicate increasing levels of disability (and dependency), and a score of 6 indicates death.
NIHSS score at Day 7 and Day 14 (or discharge if earlier) | Assessment performed at Day 7 and Day 14 (or discharge if earlier)
  The National Institutes of Health Stroke Scale to measure severity of stroke on scale 0-42.
PHE at Day 7 and Day 14 (or discharge if earlier) | Day 7 and Day 14 (or discharge if earlier)
  Perihaematomal oedema (PHE) from CT imaging data assessed at Day 7 and Day 14 (or discharge if earlier)
Total length of initial hospital stay | Within 6 months after stroke onset
  Total length of initial hospital stay within 6 months after stroke onset
Ambulatory status at hospital discharge | At the time when patient is discharged from enrolling hospital, within 6 months after stroke onset
  Assessing mobility of the patient at discharge from hospital
Place of residence at 6 months | Completed at the 6-month follow-up visit
  Assessing the patient's residence at the 6 month follow up. (example: home, rehabilitation, long term care, remains hospitalized)

CONTACTS AND LOCATIONS:
Locations (2):
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
Domain information and tabular trial results will be posted on the National Institutes of Health's website www.clinicaltrials.gov within one year of domain completion.